CLINICAL TRIAL: NCT04109638
Title: A Pilot Prospective, Randomized, Placebo-Controlled Study to Evaluate the Efficacy of Pulsed Electromagnetic Field (PEMF) Therapy in Decreasing Post-Operative Pain Following Orthopedic Surgery
Brief Title: Pulsed Electromagnetic Field (PEMF) Therapy for Post-operative Pain Following Orthopedic Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Endonovo (Unknown)
Responsible Party: Principal Investigator, Geoffrey Abrams, Assistant Professor of Orthopaedic Surgery, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 53013
Record Dates: First submitted 2019-09-27; First posted 2019-09-30 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Knee Injuries; Shoulder Injuries; Pain, Postoperative
Keywords: PEMF
MeSH Terms: conditions — Knee Injuries; Shoulder Injuries; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Active PEMF Group (Active Comparator): Participants will have a 1 in 2 chance to get the active treatment device post-operatively. The device will be attached to the post-operative dressing. The device is an Endonovo SofPulse that emits a pulsed electromagnetic field (PEMF). Single blind randomization.
  Interventions: Device: Endonovo SofPulse
- Placebo PEMF Group (Sham Comparator): Participants will have a 1 in 2 chance to get the placebo treatment device post-operatively. The device will be attached to the post-operative dressing. The Endonovo SofPulse placebo device does not emit a pulsed electromagnetic field (PEMF). Single blind randomization.
  Interventions: Device: Endonovo SofPulse

INTERVENTIONS:
Device: Endonovo SofPulse — The active device emits PEMF signal whereas the placebo device does not emit a PEMF signal. The active device is on for 15 minutes at a time, every two hours, for 10 days.
  Other Names: Endonovo tPEMF Device

SUMMARY:
The primary objective of this study is to prospectively determine, at 10 days after orthopedic shoulder or knee surgery, if pulsed electromagnetic field (PEMF) therapy is beneficial in reducing patient-reported post-operative pain, as measured by visual analog scale (VAS). The amount of pain medication taken daily and the physical function outcome scores after surgery and PEMF treatment will also be measured.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects may be male or female greater or equal to 18 years of age (≥ 18) at the time of consent.
2. Subjects who will be having shoulder or knee surgery are permitted.
3. Subject must not have used NSAIDs for one (1) week prior to surgery.

   a. a. Low-dose aspirin (81 mg) is permitted.
4. Subject must be willing and able to participate in post-operative physical therapy exercises.
5. Subject must understand and be willing to sign the IRB-approved Informed Consent Document.

Exclusion Criteria:

1. Subject has a known collagen disorder such as, but not limited to, osteogenesis imperfecta (OI) or Ehlers-Danlos syndrome (EDS).
2. Subject has a known inflammatory or autoimmune connective tissue disease such as, but not limited to, gout affecting the shoulder, scleroderma, SLE, rheumatoid disease, or calcific tendonitis of the shoulder.
3. Subject has a metabolic bone disease such as Paget's disease or osteomalacia as documented in the medical record.
4. Subject has a deltoid defect, deltoid palsy or any other pseudoparalysis.
5. Subject is diabetic.
6. Subject has HIV or hepatitis.
7. Subject has a diagnosis of fibromyalgia or other chronic pain syndrome.
8. Subject has shoulder or knee pain of unknown etiology.
9. Subject has had an active malignancy in the past 5 years OR has an active or on-going neoplastic disease, except for benign skin cancer(s).
10. Subject has undergone administration, within 30 days prior to surgery, of any type of corticosteroid (with the exception of asthma medications and ophthalmic medications), antineoplastic, immunostimulation or immunosuppressive agent.
11. Subject is septic, or has a local or systemic infection.
12. Subject has an admitted active substance abuse problem which includes recreational drugs and/or narcotics or a history of substance abuse where history is defined as "not under the care of a physician" for more than 5 years.

    a. Prescriptive medical marijuana is not permitted, including CBD oils.
13. Subject consumes more than 14 (men) or 7 (women) standard drinks (alcoholic units) per week where a drink equals a 12 oz. beer, or a 5 oz. glass of wine, or a 1.5 oz. shot of liquor.
14. Subject is currently seeking or receiving worker's compensation for this injury or for an injury that has occurred more than 12 months prior to enrollment in this study or subjects who are currently in litigation or who have a history of litigation related to musculoskeletal diagnoses.
15. Subject has major mental illnesses including major depression, bipolar disorder, schizophrenia or dementia that would prevent them from following the protocol and/or independently completing the patient reported outcomes measures.
16. Subjects who have coexistent cervical spinal pathologies such as radiculopathies or myelopathies.
17. Subject has a mental or physical condition that would prevent them from complying with the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline in pain scores on the visual analog scale (VAS) at 10 days | 10 days
  The VAS is a subjective pain scale from 0 to 10, with 0 representing no pain.

SECONDARY OUTCOMES:
Mean change from baseline in narcotic pain medicine use at 10 days | 10 days
  Pain medication will be documented every 24 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey D Abrams, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Redwood City, California, United States

IPD SHARING:
Plan to Share IPD: No